CLINICAL TRIAL: NCT02728791
Title: Comparaison de Mesure de débit Cardiaque Entre système Clearsight® et Thermodilution Transpulmonaire.
Brief Title: Comparison of Allows Measurement of Cardiac Output Between Clearsight System and Transpulmonary Thermodilution
Acronym: CONDUCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: CONDUCT (RB 15.144)
Record Dates: First submitted 2016-03-25; First posted 2016-04-05 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Shock; Cardiac Output, Low
MeSH Terms: conditions — Shock; Cardiac Output, Low

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Correlation study between the data provided by two measurement systems, trans- pulmonary thermodilution and ClearSight © (non invasive), to determine the interest in routine use (cardiac output, cardiac index, stroke volume and blood pressure).

DETAILED DESCRIPTION:
Since 2014, Edwards society has developed a completely non-invasive monitoring device for measurement of blood pressure and continuous cardiac output without inserting foreign intravascular bodies in the patient. Initially tested on healthy volunteers cardiac disease -free, the correlation with the other devices seems to be good. If this ClearSight © system show a relevant accuracy in measuring blood pressure and cardiac output with a specific ICU hospitalized population, it could justify its place in the therapeutic arsenal of monitoring in intensive care.

This is a common care ,prospective observational single center study , concerning the results of blood pressure , cardiac output values and their variations.

ELIGIBILITY:
Inclusion Criteria:

* age>18
* hospitalized in surgical ICU, with hemodynamic instability or vaso-active drugs
* No opposition formulated

Exclusion Criteria:

* Impossibility of establishment of one of the cardiac output measurement devices
* Pregnant woman
* Refuse to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients hospitalized in ICU with hemodynamic failure requiring vasoactive drugs
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-05-10 (Actual); Primary Completion 2018-12-10 (Estimated); Study Completion 2018-12-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of values and changes in cardiac index between the two devices | 2 days

SECONDARY OUTCOMES:
Comparison of values and variations in mean arterial pressure between the two devices | 2 days
Comparison of values and variations in mean cardiac output between the two devices | 2 days
Comparison of values and variations in mean stroke volume variation between the two devices | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Olivier O HUET, Principal Investigator — CHRU de Brest
Locations (1):
- CHRU BREST, Hôpital de la Cavale Blanche, Brest, France